CLINICAL TRIAL: NCT04457310
Title: A Translational and Neurocomputational Evaluation of a Dopamine Receptor 1 Partial Agonist for Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Columbia University (Other); University of Pennsylvania (Other); State University of New York Stony Brook (Unknown); Cerevel Therapeutics, LLC (Industry); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, John H. Krystal, Principal Investigator, Yale University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2000027506; 1U01MH121766-01 (NIH)
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Early Course Schizophrenia Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CVL-562 (PF-06412562) 1 mg (Experimental): Each subject will complete 5 test visits each involving the administration of CVL-562 (PF-06412562) (at different doses) or placebo. Subjects will be randomized to the order of doses of CVL-562 (PF-06412562) (1 mg, 4 mg, 15 mg, or 25 mg) or placebo for the next 5 visits. The randomization will assign 75% of patients to the highest dose on the last visit and 25% would receive the highest dose on one of the other four visits. Only the highest dose (25 mg) will be subject to this pseudo-randomization strategy; all other doses will be randomly distributed.
  Interventions: Drug: CVL-562 (PF-06412562) 1 mg
- CVL-562 (PF-06412562) 4 mg (Experimental): Each subject will complete 5 test visits each involving the administration of CVL-562 (PF-06412562) (at different doses) or placebo. Subjects will be randomized to the order of doses of CVL-562 (PF-06412562) (1 mg, 4 mg, 15 mg, or 25 mg) or placebo for the next 5 visits. The randomization will assign 75% of patients to the highest dose on the last visit and 25% would receive the highest dose on one of the other four visits. Only the highest dose (25 mg) will be subject to this pseudo-randomization strategy; all other doses will be randomly distributed.
  Interventions: Drug: CVL-562 (PF-06412562) 4 mg
- CVL-562 (PF-06412562) 15 mg (Experimental): Each subject will complete 5 test visits each involving the administration of CVL-562 (PF-06412562) (at different doses) or placebo. Subjects will be randomized to the order of doses of CVL-562 (PF-06412562) (1 mg, 4 mg, 15 mg, or 25 mg) or placebo for the next 5 visits. The randomization will assign 75% of patients to the highest dose on the last visit and 25% would receive the highest dose on one of the other four visits. Only the highest dose (25 mg) will be subject to this pseudo-randomization strategy; all other doses will be randomly distributed.
  Interventions: Drug: CVL-562 (PF-06412562) 15 mg
- CVL-562 (PF-06412562) 25 mg (Experimental): Each subject will complete 5 test visits each involving the administration of CVL-562 (PF-06412562) (at different doses) or placebo. Subjects will be randomized to the order of doses of CVL-562 (PF-06412562) (1 mg, 4 mg, 15 mg, or 25 mg) or placebo for the next 5 visits. The randomization will assign 75% of patients to the highest dose on the last visit and 25% would receive the highest dose on one of the other four visits. Only the highest dose (25 mg) will be subject to this pseudo-randomization strategy; all other doses will be randomly distributed.
  Interventions: Drug: CVL-562 (PF-06412562) 25 mg
- Placebo (Placebo Comparator): Each subject will complete 5 test visits each involving the administration of CVL-562 (PF-06412562) (at different doses) or placebo. Subjects will be randomized to the order of doses of CVL-562 (PF-06412562) (1 mg, 4 mg, 15 mg, or 25 mg) or placebo for the next 5 visits. The randomization will assign 75% of patients to the highest dose on the last visit and 25% would receive the highest dose on one of the other four visits. Only the highest dose (25 mg) will be subject to this pseudo-randomization strategy; all other doses will be randomly distributed.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CVL-562 (PF-06412562) 1 mg — Each subject will complete 5 test visits each involving the administration of CVL-562 (PF-06412562) (at different doses) or placebo. Each test visit will be separated by at least 48 hours (six half-lives of CVL-562 (PF-06412562)).
  Arms: CVL-562 (PF-06412562) 1 mg
Drug: CVL-562 (PF-06412562) 4 mg — Each subject will complete 5 test visits each involving the administration of CVL-562 (PF-06412562) (at different doses) or placebo. Each test visit will be separated by at least 48 hours (six half-lives of CVL-562 (PF-06412562)).
  Arms: CVL-562 (PF-06412562) 4 mg
Drug: CVL-562 (PF-06412562) 15 mg — Each subject will complete 5 test visits each involving the administration of CVL-562 (PF-06412562) (at different doses) or placebo. Each test visit will be separated by at least 48 hours (six half-lives of CVL-562 (PF-06412562)).
  Arms: CVL-562 (PF-06412562) 15 mg
Drug: CVL-562 (PF-06412562) 25 mg — Each subject will complete 5 test visits each involving the administration of CVL-562 (PF-06412562) (at different doses) or placebo. Each test visit will be separated by at least 48 hours (six half-lives of CVL-562 (PF-06412562)).
  Arms: CVL-562 (PF-06412562) 25 mg
Other: Placebo — Each subject will complete 5 test visits each involving the administration of CVL-562 (PF-06412562) (at different doses) or placebo. Each test visit will be separated by at least 48 hours (six half-lives of CVL-562 (PF-06412562)).
  Arms: Placebo

SUMMARY:
This study will test whether CVL-562 (PF-06412562), a dopamine 1 partial agonist novel compound, affects working memory neural circuits in patients with early episode schizophrenia. The overall aim is to establish neuroimaging biomarkers of the Dopamine Receptor 1/Dopamine Receptor 5 Family (D1R/D5R) target engagement to accelerate development of D1R/D5R agonists in humans to treat cognitive impairments that underlie functional disability in schizophrenia, a key unaddressed clinical and public health concern.

DETAILED DESCRIPTION:
This study proposes to examine the effects of CVL-562 (PF-06412562), a dopamine-1 receptor partial agonist, on the neural signal of brain regions involved in cognition in patients with schizophrenia and related psychotic disorders. The primary objective of this study is to understand the neural circuit targets of this compound as it relates to improving cognition in schizophrenia, using a spatial working memory task (sWM). The secondary objective will quantify dose-related drug effects on sWM precision based on behavioral data collected during scanning and examine effects on functional connectivity.

All patients will be psychiatrically stable with early course (psychotic symptom onset within the past 10 years) schizophrenia spectrum disorder (e.g. schizophrenia, schizoaffective disorder, or schizophreniform disorder) and will have working memory deficits (defined as below average performance on the letter n-back task of the PennCNB battery). As part of the study, they will receive oral administration of specified doses of CVL-562 (PF-06412562), in a random order with repeated functional magnetic resonance imaging and cognitive testing during those visits. The most common side effects of this compound are nausea and headache. This is a multi-site study that requires the efforts of 4 study sites in total (Columbia, State University of New York Stony Brook, UPenn, and Yale).

At time of results entry, secondary outcome results unavailable due to ongoing restrictions per the NIH

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 (including 18 years of age) and 45 (up to 45 years and 11 months) at the time of baseline study visit.
* Able to provide informed consent (as established by consent interview), and voluntary, signed informed consent prior to the performance of any study-specific procedures
* Willing and able to perform study-relevant clinical assessments and Magnetic Resonance Imaging (MRI) as assessed by research staff.
* Meet Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) criteria for schizophrenia, schizoaffective disorder, or schizophreniform disorder on the basis of the Structured Clinical Interview for DSM-5 (SCID-5).
* Be within 10 years of the onset of psychosis based on clinical assessment at the time of Visit 1.
* Treatment seeking and willing to accept the constraints on treatment entailed by the study.
* Able to demonstrate a basic ability to follow spatial working memory task instructions and perform necessary related motor functions.
* Demonstrate a premorbid IQ of ≥80 based on the Penn Reading Assessment (PRA). The PRA correlates with other measures of IQ including the Wide Range Achievement Test (WRAT), but is computerized, based in the laboratory of co-investigators Ruben C. Gur and Raquel E. Gur, and brief to administer, allowing us to lessen the assessment burden on an already lengthy first visit.
* Be fluent in English as assessed by research staff.
* Clinically stable treatment for at least two months prior to Visit 1 (no hospitalizations, or current suicidal/homicidal active ideation, intent, or plan).
* On a stable psychotropic medication regimen (can include no psychotropic medications) for at least 3 weeks prior to Visit 1, and willing to maintain an unchanged regimen during the study. If on depot antipsychotics, participants must have stable dosing for at least two consecutive injections (including the most recent one) as the most recent injections. If on Invega Trinza, there must be no plans to change dosing during the course of the study.
* For women of child bearing potential, no intention to become pregnant during the study period, and agreement to use a reliable method of birth control (e.g. Intra-Uterine Device (IUD), hormonal contraception, abstinence, condoms) during the study period. Women will be asked to continue their method of contraception for 1 month after receiving their final dose of medication. Any individual who becomes pregnant during the study will be immediately removed, and discussion of the risks and benefits of ongoing pharmacotherapy will proceed on purely clinical grounds.

Exclusion Criteria:

* Any unstable medical, psychiatric, or neurological condition (including active or otherwise remarkable suicidal or homicidal ideation) that may necessitate urgent treatment. Active medical conditions that are minor or well controlled are not exclusionary if they do not affect risk to the patient, metabolism of study drug, or the study results (e.g. well-controlled type II diabetes or hypertension) as per the judgment of the investigator.
* Be currently treated with any of the following: olanzapine, clozapine, ziprasidone or asenapine, in order to avoid prominent D1 receptor effects.
* Any major neurological disease, brain injury, epilepsy, or history of severe head trauma, including concussion with loss of consciousness greater than or equal to > 15 minutes, or of psychosurgery.
* History of significant cardiac disease (ex: ischemia, arrhythmia).
* Any clinically significant abnormality on baseline medical screening tests (electrocardiogram (EKG), complete blood count with differential (CBC), complete metabolic profile (CMP).
* Hepatitis B or C (by report or testing) in the presence of abnormal liver function tests
* Human Immunodeficiency Virus (HIV) or Acquired Immune Deficiency Syndrome (AIDS) (by report or by testing) due cognitive effects of HIV and AIDS.
* Baseline EKG showing prolonged QTc interval (>450 for males, >470 for females, Framingham correction(3)), with repeat measurement showing the same abnormality.
* Current mood episode meeting criteria for a major depressive episode or a manic or hypomanic episode.
* History of electroconvulsive therapy (ECT) or treatment with neurostimulation in the past 6 months, or with plans to begin either such treatment during the study.
* History of ADHD pre-morbid to the onset of psychosis or other psychiatric illnesses that may be accompanied by cognitive impairments.
* Meeting SCID-5 moderate or severe substance use disorder for any substance other than nicotine within the 3 months prior to the initial assessment.
* Positive urine toxicology testing for any substance other than marijuana or those prescribed for medical reasons at Visits 1-6.
* Pregnancy or intention to become pregnant during the study.
* Lactating/breast-feeding or intending to do so during the study
* Any non-MRI compatible metal in the body or other contraindication to MR imaging. A copper IUD is allowable if permitted by local MRI practices.
* Severe claustrophobia, back pain, morbid obesity, or other condition that may make an extended MR session difficult or lead to excessive movement during the imaging session.
* Color blindness, strabismus or other uncorrectable visual problems. Those wearing glasses would be asked to use MRI-safe glasses.
* Daily use of the following medication within 10 days prior to the initial visit or during the study: Long-acting nighttime or daytime gamma aminobutyric acid-A (GABA-A) receptor facilitators; anticonvulsant medications used at high doses or for seizure control, or psychostimulants or medical cannabis. Participants can be re-assessed for eligibility once they have been free of daily use of these medications for >10 days. Participants may take non-GABAergic sleep medications, short-acting GABA receptor facilitators (benzodiazepine, non-benzodiazepine) prior to and during the study.
* Any change in type or dose of psychotropic medications within 3 weeks prior to initial visit or during study to avoid transient effects of medication regimen change. Medication type and dose will be carefully recorded and used as a covariate in analyses. Participants can be re-assessed for eligibility once they have been on a stable dose of medication for >3 weeks.
* CVL-562 is metabolized by P450 CYP3A4. In order to avoid pharmacokinetic interactions, medications or substances that induce (barbiturate, carbamazepine, etc.) or are moderate-strong inhibitors (ketoconazole, etc.; grapefruit juice) are excluded if used within 10 days prior to or during study. Participants can be re-assessed for eligibility once they have been free of these medications/substances for >10 days.
* Active attempts to discontinue smoking, vaping or other nicotine products within the 3 weeks prior to study or during the study. Participants can be re-assessed once quit attempt is stable.
* Diastolic blood pressure >95 or <50 mmHg or systolic blood pressure > 170 or <80 mmHg with repeat measurement showing the same abnormality.
* History of allergy or other contraindication to the proposed pharmacotherapy.
* Other medication treatment with which proposed pharmacotherapy is contraindicated, in the opinion of study psychiatrists or of a subject's prescribing psychiatrist.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Krystal, MD, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Yale University, New Haven, Connecticut
  - Columbia University, New York, New York
  - Stony Brook University, Stony Brook, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made publicly available through the NIMH Data Archive (NDAR) with data uploaded every 6 months.
Time Frame: Six months after publication.
Access Criteria: All neuroimaging data will be shared through the National Institute of Mental Health Data Archive (NDA). All requests for accessing these data will be reviewed by the National Institute of Mental Health.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data for participants who started test visits at Columbia was required to be removed due to research restrictions per the NIH (see GCE). Secondary outcome results unavailable due to ongoing restrictions per the NIH.
Groups:
- All Study Participants: Each subject will complete 5 test visits each involving the administration of CVL-562 (PF-06412562) (at different doses) or placebo. All participants will receive all doses (a different dose at each of the 5 visits.)
Period: Overall Study
Arm/Group | All Study Participants
Started | 112
Have MRI Data | 52
Usable Full MRI Data (Analysis Population) (Only full usable MRI data can be analyzed. Participants without full usable MRI data (missing scans, incomplete scans, etc) cannot be analyzed.) | 50
Participants Started at Columbia Site | 28
Participants Started at All Other Sites (Demographic and Adverse Event results available.) | 84
Received CVL-562 (PF-06412562) 1 mg | 78
Received CVL-562 (PF-06412562) 4 mg | 77
Received CVL-562 (PF-06412562) 15 mg | 75
Received CVL-562 (PF-06412562) 25 mg | 70
Received Placebo | 77
Completed (Attended every test visit) | 71
Not Completed | 41

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are provided for the 84 participants with available data.
Arm/Group | All Study Participants
Number analyzed (Participants) | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.06 (5.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 28
  White | 29
  More than one race | 18
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 84

OUTCOME MEASURES:

1. Primary Outcome: Neural Activity Across Brain Regions During a Spatial Working Memory (sWM) Task- Condition 2
Description: Neural activity will be measured by blood oxygen level dependent (BOLD) signal that will be assessed during functional magnetic resonance (fMRI) sessions. During each fMRI session, subjects will participate in a sWM task that involves the ability to keep a spatial location in mind over a short period of time. The sWM task includes four conditions: 1) only sWM; 2) a motor response without sWM; 3) sWM with a distracter presented near the original memory location; and 4) sWM with a distractor presented far away from the original memory location. For each condition, BOLD signal will be assessed over 20 timepoints, each measuring for 0.8 seconds [total 16s]. Each subject will undergo 5 fMRI sessions, one at each dose.
Time Frame: Up to two hours for each fMRI session
Measure: Mean (Standard Deviation); unit: percentage signal change
Arm/Group | CVL-562 (PF-06412562) 1 mg | CVL-562 (PF-06412562) 4 mg | CVL-562 (PF-06412562) 15 mg | CVL-562 (PF-06412562) 25 mg | Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50
percentage signal change
  Second 0.8 | -0.076 (0.165) | -0.090 (0.177) | -0.072 (0.180) | -0.136 (0.169) | -0.064 (0.161)
  Second 1.6 | -0.090 (0.217) | -0.097 (0.225) | -0.083 (0.223) | -0.167 (0.207) | -0.067 (0.212)
  Second 2.4 | -0.045 (0.235) | -0.042 (0.231) | -0.039 (0.235) | -0.135 (0.213) | -0.043 (0.232)
  Second 3.2 | 0.024 (0.238) | 0.028 (0.239) | 0.031 (0.245) | -0.066 (0.228) | 0.020 (0.223)
  Second 4.0 | 0.092 (0.240) | 0.094 (0.256) | 0.104 (0.246) | -0.012 (0.235) | 0.072 (0.237)
  Second 4.8 | 0.119 (0.261) | 0.137 (0.259) | 0.143 (0.257) | 0.027 (0.251) | 0.110 (0.248)
  Second 5.6 | 0.105 (0.271) | 0.144 (0.263) | 0.153 (0.265) | 0.033 (0.246) | 0.113 (0.246)
  Second 6.4 | 0.078 (0.280) | 0.118 (0.256) | 0.127 (0.260) | 0.006 (0.243) | 0.100 (0.257)
  Second 7.2 | 0.038 (0.287) | 0.097 (0.257) | 0.086 (0.251) | -0.028 (0.239) | 0.061 (0.254)
  Second 8.0 | -0.009 (0.294) | 0.064 (0.260) | 0.055 (0.238) | -0.059 (0.228) | 0.025 (0.259)
  Second 8.8 | -0.036 (0.292) | 0.045 (0.248) | 0.020 (0.227) | -0.087 (0.220) | 0.001 (0.262)
  Second 9.6 | -0.045 (0.288) | 0.032 (0.242) | -0.007 (0.230) | -0.091 (0.207) | -0.020 (0.247)
  Second 10.4 | -0.054 (0.289) | 0.027 (0.235) | -0.015 (0.237) | -0.093 (0.209) | -0.030 (0.253)
  Second 11.2 | -0.049 (0.292) | 0.036 (0.237) | -0.012 (0.232) | -0.092 (0.212) | -0.038 (0.248)
  Second 12.0 | -0.025 (0.289) | 0.051 (0.250) | -0.005 (0.240) | -0.073 (0.216) | -0.034 (0.258)
  Second 12.8 | -0.017 (0.275) | 0.049 (0.243) | 0.003 (0.247) | -0.052 (0.216) | -0.033 (0.262)
  Second 13.6 | 0.015 (0.275) | 0.072 (0.238) | 0.033 (0.257) | -0.025 (0.214) | -0.004 (0.271)
  Second 14.4 | 0.073 (0.278) | 0.124 (0.242) | 0.083 (0.269) | 0.028 (0.223) | 0.056 (0.281)
  Second 15.2 | 0.138 (0.281) | 0.177 (0.248) | 0.153 (0.288) | 0.091 (0.238) | 0.127 (0.287)
  Second 16.0 | 0.187 (0.290) | 0.229 (0.251) | 0.225 (0.310) | 0.130 (0.277) | 0.175 (0.297)

2. Secondary Outcome: Performance During Spatial Working Memory (sWM) Task
Description: During each fMRI session, subjects will participate in a sWM task that involves the ability to keep a spatial location in mind over a short period of time. The sWM task includes four conditions: 1) only sWM; 2) a motor response without sWM; 3) sWM with a distracter presented near the original memory location; and 4) sWM with a distractor presented far away from the original memory location. Performance will be assessed with the average accuracy measured during this task for each task condition and each CVL-562 (PF-06412562) dose. Accuracy refers to the angular distance between a cued location and a participant's memory of the location. The range of accuracy is between 0-180 degrees. 0 degrees would indicate the best possible performance, and 180 degrees the worst performance. Each subject will undergo 5 fMRI sessions, each at a different dose of CVL-562 (PF-06412562).
Time Frame: Up to two hours for each fMRI session.
Reporting Status: Not Posted

3. Secondary Outcome: Association Between Neural Activity and Task Performance
Description: Neural activity will be measured by blood oxygen level dependent (BOLD) signal that will be assessed during fMRI, where subjects will participate in a spatial working memory (sWM) task. The sWM includes four conditions: 1) only sWM; 2) a motor response without sWM; 3) sWM with a distracter presented near the original memory location; and 4) sWM with a distractor presented far away from the original memory location. The performance of sWM at each trial of each condition will be used as the predictor variable, and the BOLD signal at the corresponding trial and condition will be used as the outcome variable. A trial refers to a single probing and measurement of sWM, and is repeatedly presented to get a number of sWM measurements. The performance of sWM from each trial will be regressed with the BOLD signal from that trial, and we will report the resulting beta weights at each condition and dose. Each subject will undergo 5 fMRI sessions, each at a different dose of CVL-562 (PF-06412562).
Time Frame: Up to two hours for each fMRI session.
Reporting Status: Not Posted

4. Secondary Outcome: Functional Connectivity Across Brain Regions With the Fronto-parietal Network During sWM Task
Description: Functional connectivity will be assessed during each fMRI session. Functional connectivity refers to the correlation between the time series of different brain regions collected during fMRI. During each fMRI session, subjects will participate in a sWM task that involves the ability to keep a spatial location in mind over a short period of time. The sWM task includes four conditions: 1) only sWM; 2) a motor response without sWM; 3) sWM with a distracter presented near the original memory location; and 4) sWM with a distractor presented far away from the original memory location. For each condition, the functional connectivity of the fronto-parietal network will be measured with the rest of the brain. The range of functional connectivity is between -4.95 and 4.95. -4.95 would indicate highly negative functional connectivity and 4.95 would indicate highly positive functional connectivity. Each subject will undergo 5 fMRI sessions, each at a different dose of CVL-562 (PF-06412562).
Time Frame: Up to two hours for each fMRI session.
Reporting Status: Not Posted

5. Secondary Outcome: Resting State Global Brain Functional Connectivity
Description: BOLD signal will be collected during the resting state aspect of the fMRI session, using a data-driven global brain connectivity (GBC) metric. GBC examines connectivity from a given voxel (or area) to all other voxels (or areas) simultaneously by computing average connectivity strength. The range of GBC is between -4.95 and 4.95. -4.95 would indicate highly negative broad functional connectivity in synchrony with the rest of the brain and 4.95 would indicate highly positive broad functional connectivity in synchrony with the rest of the brain. GBC will be obtained at each PF-06412562 dose.
Time Frame: Up to two hours for each fMRI session.
Reporting Status: Not Posted

6. Secondary Outcome: Proportion of Participants With Change in Blood Oxygen Level Dependent (BOLD) Signal During Spatial Working Memory (sWM) Task.
Description: The dose-response in BOLD signal will be examined for each individual participant to see how many participants exhibit a change in BOLD signal overall. For each individual, binary outcome will be calculated based on a Dose by Condition by Time within subject analysis of BOLD signal. We will report the proportion of participants that exhibits a dose response.
Time Frame: Up to two hours for each fMRI session.
Reporting Status: Not Posted

7. Secondary Outcome: Spatial Similarity of Resting State Global Brain Functional Connectivity With Transcriptomic Maps.
Description: Transcriptomics maps will be derived from the Allen Human Brain Atlas (AHBA), which provides gene expression data mapped to the cortical surface. The spatial similarity of resting state global brain functional connectivity (GBC) and gene expression patterns for the D1/D5 receptors will be assessed for each CVL-562 (PF-06412562) dose. The spatial similarity refers to correlation between GBC maps and the cortical gene expression maps. Each subject will undergo 5 fMRI sessions, each at a different dose of CVL-562 (PF-06412562).
Time Frame: Up to two hours for each fMRI session.
Reporting Status: Not Posted

8. Primary Outcome: Neural Activity Across Brain Regions During a Spatial Working Memory (sWM) Task- Condition 1
Description: as for outcome 1
Time Frame: Up to two hours for each fMRI session
Measure: Mean (Standard Deviation); unit: percentage signal change
Arm/Group | CVL-562 (PF-06412562) 1 mg | CVL-562 (PF-06412562) 4 mg | CVL-562 (PF-06412562) 15 mg | CVL-562 (PF-06412562) 25 mg | Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50
percentage signal change
  Second 0.8 | -0.070 (0.155) | -0.040 (0.148) | -0.060 (0.164) | -0.065 (0.151) | -0.081 (0.152)
  Second 1.6 | -0.086 (0.200) | -0.036 (0.197) | -0.076 (0.218) | -0.079 (0.184) | -0.093 (0.187)
  Second 2.4 | -0.042 (0.200) | 0.013 (0.214) | -0.039 (0.216) | -0.045 (0.197) | -0.053 (0.198)
  Second 3.2 | 0.025 (0.228) | 0.074 (0.225) | 0.025 (0.220) | 0.010 (0.193) | 0.012 (0.204)
  Second 4.0 | 0.071 (0.243) | 0.131 (0.223) | 0.081 (0.245) | 0.060 (0.207) | 0.068 (0.216)
  Second 4.8 | 0.089 (0.243) | 0.151 (0.223) | 0.109 (0.266) | 0.091 (0.224) | 0.098 (0.224)
  Second 5.6 | 0.087 (0.251) | 0.145 (0.219) | 0.096 (0.287) | 0.089 (0.228) | 0.090 (0.228)
  Second 6.4 | 0.054 (0.255) | 0.126 (0.212) | 0.067 (0.280) | 0.067 (0.236) | 0.059 (0.237)
  Second 7.2 | 0.011 (0.250) | 0.088 (0.213) | 0.032 (0.279) | 0.040 (0.238) | 0.032 (0.245)
  Second 8.0 | -0.013 (0.254) | 0.056 (0.207) | -0.009 (0.273) | 0.019 (0.243) | 0.000 (0.240)
  Second 8.8 | -0.038 (0.256) | 0.043 (0.216) | -0.033 (0.269) | -0.010 (0.228) | -0.018 (0.242)
  Second 9.6 | -0.056 (0.258) | 0.027 (0.223) | -0.038 (0.265) | -0.022 (0.223) | -0.042 (0.246)
  Second 10.4 | -0.068 (0.246) | 0.024 (0.214) | -0.032 (0.267) | -0.031 (0.216) | -0.042 (0.237)
  Second 11.2 | -0.053 (0.233) | 0.028 (0.210) | -0.024 (0.267) | -0.038 (0.206) | -0.044 (0.233)
  Second 12.0 | -0.041 (0.235) | 0.032 (0.211) | 0.000 (0.269) | -0.040 (0.229) | -0.038 (0.235)
  Second 12.8 | -0.026 (0.241) | 0.037 (0.227) | 0.005 (0.272) | -0.029 (0.217) | -0.029 (0.236)
  Second 13.6 | 0.014 (0.246) | 0.077 (0.231) | 0.046 (0.273) | 0.002 (0.222) | 0.019 (0.242)
  Second 14.4 | 0.079 (0.251) | 0.142 (0.234) | 0.101 (0.281) | 0.056 (0.235) | 0.086 (0.249)
  Second 15.2 | 0.146 (0.279) | 0.203 (0.246) | 0.165 (0.290) | 0.134 (0.246) | 0.150 (0.269)
  Second 16.0 | 0.200 (0.286) | 0.247 (0.265) | 0.209 (0.307) | 0.172 (0.258) | 0.204 (0.287)

9. Primary Outcome: Neural Activity Across Brain Regions During a Spatial Working Memory (sWM) Task- Condition 3
Description: as for outcome 1
Time Frame: Up to two hours for each fMRI session
Measure: Mean (Standard Deviation); unit: percentage signal change
Arm/Group | CVL-562 (PF-06412562) 1 mg | CVL-562 (PF-06412562) 4 mg | CVL-562 (PF-06412562) 15 mg | CVL-562 (PF-06412562) 25 mg | Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50
percentage signal change
  Second 0.8 | -0.108 (0.134) | -0.100 (0.112) | -0.122 (0.130) | -0.072 (0.119) | -0.122 (0.095)
  Second 1.6 | -0.108 (0.150) | -0.116 (0.118) | -0.129 (0.137) | -0.077 (0.127) | -0.128 (0.105)
  Second 2.4 | -0.063 (0.153) | -0.072 (0.122) | -0.073 (0.137) | -0.043 (0.127) | -0.078 (0.099)
  Second 3.2 | 0.017 (0.147) | -0.004 (0.122) | -0.003 (0.131) | 0.025 (0.121) | 0.004 (0.111)
  Second 4.0 | 0.074 (0.151) | 0.044 (0.134) | 0.053 (0.127) | 0.069 (0.114) | 0.054 (0.116)
  Second 4.8 | 0.108 (0.145) | 0.067 (0.134) | 0.087 (0.129) | 0.102 (0.105) | 0.074 (0.116)
  Second 5.6 | 0.100 (0.162) | 0.072 (0.120) | 0.095 (0.128) | 0.095 (0.110) | 0.070 (0.115)
  Second 6.4 | 0.086 (0.167) | 0.051 (0.122) | 0.079 (0.126) | 0.058 (0.109) | 0.046 (0.110)
  Second 7.2 | 0.062 (0.171) | 0.035 (0.132) | 0.059 (0.111) | 0.040 (0.104) | 0.033 (0.110)
  Second 8.0 | 0.052 (0.159) | 0.042 (0.128) | 0.059 (0.111) | 0.048 (0.098) | 0.037 (0.103)
  Second 8.8 | 0.084 (0.145) | 0.083 (0.143) | 0.095 (0.113) | 0.089 (0.104) | 0.074 (0.098)
  Second 9.6 | 0.127 (0.146) | 0.119 (0.147) | 0.128 (0.109) | 0.125 (0.113) | 0.115 (0.109)
  Second 10.4 | 0.158 (0.140) | 0.130 (0.136) | 0.126 (0.109) | 0.147 (0.127) | 0.141 (0.119)
  Second 11.2 | 0.161 (0.141) | 0.125 (0.144) | 0.116 (0.128) | 0.139 (0.137) | 0.144 (0.119)
  Second 12.0 | 0.136 (0.141) | 0.094 (0.153) | 0.094 (0.123) | 0.117 (0.142) | 0.117 (0.125)
  Second 12.8 | 0.107 (0.147) | 0.057 (0.149) | 0.063 (0.113) | 0.085 (0.130) | 0.086 (0.129)
  Second 13.6 | 0.091 (0.137) | 0.049 (0.137) | 0.042 (0.114) | 0.077 (0.125) | 0.077 (0.134)
  Second 14.4 | 0.116 (0.135) | 0.065 (0.140) | 0.068 (0.118) | 0.094 (0.134) | 0.098 (0.140)
  Second 15.2 | 0.148 (0.145) | 0.095 (0.162) | 0.108 (0.141) | 0.129 (0.142) | 0.138 (0.150)
  Second 16.0 | 0.180 (0.182) | 0.131 (0.171) | 0.165 (0.164) | 0.169 (0.156) | 0.181 (0.160)

10. Primary Outcome: Neural Activity Across Brain Regions During a Spatial Working Memory (sWM) Task- Condition 4
Description: as for outcome 1
Time Frame: Up to two hours for each fMRI session
Measure: Mean (Standard Deviation); unit: percentage signal change
Arm/Group | CVL-562 (PF-06412562) 1 mg | CVL-562 (PF-06412562) 4 mg | CVL-562 (PF-06412562) 15 mg | CVL-562 (PF-06412562) 25 mg | Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50
percentage signal change
  Second 0.8 | -0.124 (0.119) | -0.120 (0.134) | -0.133 (0.118) | -0.137 (0.109) | -0.110 (0.124)
  Second 1.6 | -0.120 (0.133) | -0.123 (0.144) | -0.138 (0.132) | -0.146 (0.113) | -0.109 (0.137)
  Second 2.4 | -0.079 (0.139) | -0.090 (0.134) | -0.090 (0.137) | -0.109 (0.113) | -0.066 (0.140)
  Second 3.2 | -0.021 (0.139) | -0.023 (0.137) | -0.022 (0.124) | -0.040 (0.111) | -0.013 (0.133)
  Second 4.0 | 0.043 (0.142) | 0.034 (0.138) | 0.044 (0.124) | 0.011 (0.119) | 0.046 (0.131)
  Second 4.8 | 0.078 (0.143) | 0.060 (0.136) | 0.079 (0.118) | 0.039 (0.138) | 0.079 (0.134)
  Second 5.6 | 0.085 (0.144) | 0.050 (0.135) | 0.093 (0.118) | 0.049 (0.146) | 0.062 (0.118)
  Second 6.4 | 0.068 (0.141) | 0.028 (0.140) | 0.078 (0.131) | 0.039 (0.139) | 0.044 (0.109)
  Second 7.2 | 0.048 (0.141) | 0.017 (0.147) | 0.051 (0.133) | 0.010 (0.142) | 0.021 (0.106)
  Second 8.0 | 0.046 (0.129) | 0.033 (0.146) | 0.048 (0.131) | 0.026 (0.131) | 0.026 (0.094)
  Second 8.8 | 0.066 (0.127) | 0.085 (0.150) | 0.073 (0.123) | 0.043 (0.136) | 0.041 (0.093)
  Second 9.6 | 0.090 (0.137) | 0.109 (0.143) | 0.101 (0.115) | 0.077 (0.144) | 0.071 (0.097)
  Second 10.4 | 0.096 (0.143) | 0.125 (0.137) | 0.115 (0.120) | 0.085 (0.135) | 0.079 (0.111)
  Second 11.2 | 0.084 (0.148) | 0.118 (0.131) | 0.097 (0.116) | 0.067 (0.131) | 0.070 (0.110)
  Second 12.0 | 0.060 (0.145) | 0.084 (0.126) | 0.073 (0.120) | 0.052 (0.133) | 0.062 (0.120)
  Second 12.8 | 0.026 (0.163) | 0.053 (0.129) | 0.047 (0.128) | 0.025 (0.123) | 0.033 (0.123)
  Second 13.6 | 0.010 (0.150) | 0.037 (0.121) | 0.046 (0.135) | 0.003 (0.118) | 0.021 (0.128)
  Second 14.4 | 0.042 (0.158) | 0.058 (0.118) | 0.089 (0.151) | 0.033 (0.125) | 0.049 (0.134)
  Second 15.2 | 0.074 (0.169) | 0.095 (0.138) | 0.129 (0.172) | 0.059 (0.148) | 0.086 (0.142)
  Second 16.0 | 0.118 (0.161) | 0.122 (0.148) | 0.172 (0.154) | 0.091 (0.190) | 0.120 (0.144)

ADVERSE EVENTS:
Time Frame: 21 weeks
Groups:
- CVL-562 (PF-06412562) 1mg: All subjects received 1mg CVL-562 (PF-06412562)
- CVL-562 (PF-06412562) 4mg: All subjects received 4mg CVL-562 (PF-06412562)
- CVL-562 (PF-06412562) 15mg: All subjects received 15mg CVL-562 (PF-06412562)
- CVL-562 (PF-06412562) 25mg: All subjects received 25mg CVL-562 (PF-06412562)
- Placebo: All subjects received Placebo
- Adverse Event Prior to Starting Intervention: Adverse event occurred prior to starting intervention
Arm/Group | CVL-562 (PF-06412562) 1mg | CVL-562 (PF-06412562) 4mg | CVL-562 (PF-06412562) 15mg | CVL-562 (PF-06412562) 25mg | Placebo | Adverse Event Prior to Starting Intervention
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/84 | 0/84 | 0/84 | 0/84 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/84 | 1/84 | 0/84 | 0/84 | 1/84
Other Adverse Events (participants affected / at risk) | 20/84 | 21/84 | 29/84 | 35/84 | 24/84 | 0/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CVL-562 (PF-06412562) 1mg (N=84) | CVL-562 (PF-06412562) 4mg (N=84) | CVL-562 (PF-06412562) 15mg (N=84) | CVL-562 (PF-06412562) 25mg (N=84) | Placebo (N=84) | Adverse Event Prior to Starting Intervention (N=84)
worsening pyschosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
worsening pyschosis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
fall and loss of vision in eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CVL-562 (PF-06412562) 1mg (N=84) | CVL-562 (PF-06412562) 4mg (N=84) | CVL-562 (PF-06412562) 15mg (N=84) | CVL-562 (PF-06412562) 25mg (N=84) | Placebo (N=84) | Adverse Event Prior to Starting Intervention (N=84)
sleepiness (Nervous system disorders) | 20 | 21 | 29 | 21 | 24 | NA
nausea (Gastrointestinal disorders) | 5 | 6 | 16 | 35 | 3 | NA
headache (Nervous system disorders) | 8 | 8 | 12 | 14 | 6 | NA
low energy (General disorders) | 8 | 5 | 4 | 11 | 11 | NA
light-headedness (Nervous system disorders) | 7 | 7 | 10 | 10 | 7 | NA
anxiety (Psychiatric disorders) | 7 | 6 | 4 | 7 | 3 | NA
abdominal discomfort (Gastrointestinal disorders) | 3 | 2 | 6 | 4 | 6 | NA
vomiting (General disorders) | 0 | 1 | 3 | 14 | 0 | NA
worsened psychosis (Psychiatric disorders) | 3 | 2 | 5 | 5 | 4 | NA
Back pain (Nervous system disorders) | 0 | 2 | 2 | 1 | 2 | NA

LIMITATIONS AND CAVEATS:
Secondary outcome data is unavailable at this time due to the ongoing restrictions at the Columbia/New York State Psychiatric Institute (NYSPI) site, preventing data access and sharing described in the approved GCE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT04457310/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT04457310/ICF_001.pdf